CLINICAL TRIAL: NCT01666938
Title: The Use of a Telephone Counselling as a Strategy to Promote Physical Activity in Diabetes Mellitus People
Brief Title: Telephone Counselling to Promote Physical Activity in Diabetes Mellitus People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Gabriel Guidorizzi Zanetti, Principal Investigator, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CSE-1410/2011
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2013-03

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Telephone; Physical activity
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity

ARMS (2):
- Diabetes Education Group & Telephone counseling (Experimental): This step was done for four months.
  Interventions: Other: Diabetes Education Group; Other: Telephone Counseling
- Telephone counseling about physical activity (Active Comparator): This step was done for four months.
  Interventions: Other: Telephone Counseling

INTERVENTIONS:
Other: Diabetes Education Group — Diabetes Education Group: Diabetes Education for four month, one time per week.
  Arms: Diabetes Education Group & Telephone counseling
Other: Telephone Counseling — Telephone counseling: 12 phone calls for four months about physical activity. During the first and second month, was done four phone calls each month. During the third and fourth month, was done two phone calls per month.

SUMMARY:
The purpose of this study is to investigate the effects of phone counselling support as a strategy to increase physical activity in people with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 2 diabetes mellitus
* age between 18 and 80 years
* both sexes
* medical recommendation for physical activity
* ability to listen and answer questions
* have cell phone and/or residential
* be registered the Center for Family Health 03 in 2012
* People should also produce higher frequency than 75% stake in the proposed activities Diabetes Education Group and telephone counseling

Exclusion Criteria: People who do not attend the criteria for inclusion.

* did not have clinical diagnosis of type 2 diabetes mellitus
* did not have age between 18 and 80 years
* did not have medical recommendation for physical activity
* did not have ability to listen and answer questions
* did not have cell phone and/or residential
* do not be registered the Center for Family Health 03 in 2012
* People who did not participate in 75% of the activities of the Group proposed the Diabetes Education and telephone counseling

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-04; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
level of physical activity | four months
  It was used the international physical activity questionnaire (IPAQ) to classify the level of physical activity

SECONDARY OUTCOMES:
Metabolic Control | Four Months
  * Body Mass Index
  * Waist Circumference
  * Mean Systolic Blood Pressure
  * Mean Diastolic Blood Pressure
  * Fasting Glucose
  * Low Density Lipoprotein (LDL)
  * High Density Lipoprotein
  * Total Cholesterol
  * Triglycerides
  * Glycated Hemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Guidorizzi Zanetti, graduated, Principal Investigator — University of Sao Paulo
Locations (1):
- Center for Family Health 03, Ribeirão Preto, São Paulo, Brazil